CLINICAL TRIAL: NCT04132154
Title: Prevention of Hypothermia During Caesarean Section: Forced-air Warming and Continuous Core Temperature Monitoring With Zero-heat-flux
Brief Title: Prevention of Hypothermia During Caesarean Section: Continuous Core Temperature Monitoring With Zero-heat-flux
Status: Completed | Type: Observational
Sponsor: St. Marien-Hospital Düren (Other)
Collaborators: Institute for Occupational, Social and Environmental Medicine, RWTH Aachen University (Unknown); Department of Anaesthesiology and Intensive Care Medicine, Hospital Düren (Unknown)
Responsible Party: Principal Investigator, Laurentiu Marin, MD, Anaesthesiologist, St. Marien-Hospital Düren
Other Study IDs: SMHDN012019
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Inadvertent Perioperative Hypothermia
Keywords: cesarean section; C-Section; Hypothermia; Spinal Anesthesia; caesarean section; zero heat flux technology; active warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Warming: Patients in this group were treated according to our institution's old protocol and did not receive any warming intervention during the surgical procedure.
- Active Warming: This group will include the patients treated after the implementation of the S3 Guidelines for prevention of hypothermia. For this purpose convective warming through an underbody blanket was used during the surgical procedure
  Interventions: Procedure: Convective Forced-Air Active Warming

INTERVENTIONS:
Procedure: Convective Forced-Air Active Warming — Underbody Blanket Model 585 of the 3M BairHugger Series
  Groups: Active Warming

SUMMARY:
Nowadays, caesarean sections account for about 7% of all surgical procedures worldwide. Over 30% of the patients undergoing a caesarean section experience a fall of the body core temperature under 36°C during the procedure. Following a retrospective cohort design, this study aims to examine the magnitude of hypothermia in the parturient and newborn population as well as the impact and efficiency of forced-air warming on preventing it. The researchers plan to conduct a retrospective analysis of the caesarean section treatment protocol at our institution over a period of 5 months including approximately 300 patients who underwent both elective and emergency caesarean sections.

DETAILED DESCRIPTION:
This research seeks to address the necessity of standardizing the use of forced-air warming and monitoring the maternal temperature during caesarean sections. We will also examine the impact of the maternal hypothermia on the newborn temperatures at the time of partus and also 2 hours after birth. The key research question of this study is whether the use of forced-air warming will significantly lower the hypothermia rates and account for a faster temperature recovery in our parturient patients.

A major contribution of our research is that it provides modern high-resolution, continuous and user-error free thermometry. This is achieved through zero-heat-flux technology and automatically recorded by data-loggers. Also, the heterogeneity of our study population, which has not been attended in previous studies, corresponds to the clinical reality of the most obstetric clinics.

This research could provide new information about the necessity of standardizing the use of forced-air warming and monitoring the maternal temperature during caesarean sections, in the concept of bonding the babies to the mother's chest immediately after birth, and derive practical implications on the efficiency of intraoperative warming for the standard clinical routine of the majority of the obstetric clinics.

ELIGIBILITY:
Inclusion Criteria:

Included will be all Caesarean section deliveries under spinal anaesthesia at our facility in the period from 01.04.2019 to 31.08.2019

Exclusion Criteria:

* different anaesthesia procedure (e.g. intubation anaesthesia, peridural anaesthesia etc.),
* American Society of Anesthesiologists (ASA) Classification III or higher,
* BMI( Body mass index) >45 kg·m-2,
* patients with incomplete documentation,
* estimated perioperative blood loss > 500ml,
* other perioperative complications (ex. insufficient analgesia and change of anaesthesia procedure).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Included will be patients undergoing spinal anaesthesia for elective and emergency caesarean delivery in accordance with our clinical day-to-day operative protocol.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Hypothermia rate OR | Through completion of the surgical procedure, an average of 1 hour
  Hypothermia rate in % intraoperatively. The temperature measurements will be started prior to the induction of the anaesthesia and ended when the patient leaves the OR (operating room).
Hypothermia rate RR | Through completion of the postoperative recovery, an average of 2 hours
  Hypothermia rate in % in the RR (recovery room). The temperature measurements will be started when the patient enters the RR and ended approximately after 2-3 hours when the patient leaves the RR

SECONDARY OUTCOMES:
Delta_Temp | Through completion of the surgical procedure, an average of 1 hour
  Temp= Temperature. Delta_Temp=The difference between Tmax -Tmin( the maximum and the minimum recorded temperatures)
Delta_Time | Through completion of the surgical procedure, an average of 1 hour
  The time from the induction of anesthesia to Nadir of temperature values
Delta_recovery | Through completion of the surgical procedure and the postoperative recovery phase , an average of 3 hour
  The time from Tmin (minimum recorded temperature values) to the recovery of 30% of the dropped body core temperature in degrees Celsius.

OTHER OUTCOMES:
Newborn pH | At birth
  For pH values only samples of umbilical venous blood will be used. point-of-care arterial-blood gas (ABG) devices will be used for testing the samples.
Newborn BE | At birth
  For BE (Base excess) values only samples of umbilical venous blood will be used. point-of-care arterial-blood gas (ABG) devices will be used for testing the samples.
Newborn APGAR score | At 1, 5 and 10 minutes after birth
  The international standard APGAR Score will be asserted at 1, 5 and 10 minutes after birth. The minimum score is 0 and the maximum 10, a greater score meaning a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Laurentiu Marin, MD, Principal Investigator — Anaesthesiologist
Locations (1):
- St. Marien Hospital, Düren, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
no IPD sharing